CLINICAL TRIAL: NCT02178345
Title: Predictive MRI Metrics for Tumor Aggressiveness in Papillary Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-126
Record Dates: First submitted 2014-06-25; First posted 2014-06-30 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Papillary Thyroid Cancer
Keywords: MRI; 14-126
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Magnetic Resonance Spectroscopy; delta 24-sterol reductase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Surgical patients: The patients will undergo DW-MRI and (if patient is eligible and agrees) DCE-MRI study prior to surgery. The maximum time interval allowed between the MRI study and surgery will be six months.
  Interventions: Procedure: diffusion weighted (DW) MRI; Procedure: dynamic contrast agent (DCE) MRI
- surveillance management patients: The patients will undergo DW-MRI and (if patient is eligible and agrees) DCE-MRI study while being on active surveillance.These patients can also receive the same DW and DCE MRI as a followup a year after the first.
  Interventions: Procedure: diffusion weighted (DW) MRI; Procedure: dynamic contrast agent (DCE) MRI

INTERVENTIONS:
Procedure: diffusion weighted (DW) MRI
Procedure: dynamic contrast agent (DCE) MRI

SUMMARY:
Magnetic resonance imaging (MRI) is a diagnostic technique that takes pictures of organs of the body. It uses magnetic fields and radio waves that cannot be felt. Perfusion MRI uses faster imaging. It also includes a contrast material that is given by vein. This makes specific organs, blood vessels, or tumors easier to see. Diffusion MRI lets us measure the motion of water in the tumor.

Perfusion and diffusion MRI give extra information which is not available with the regular MRI. A regular MRI only shows pictures of the tumor. Thyroid MRI scans are not part of the current standard of care. The purpose of this study is to see if new MRI methods can give us more information about the tumor.

DETAILED DESCRIPTION:
The aim of this pilot study clinical trial is to provide MRI biomarkers as quantitative (surrogate) biomarkers of aggressiveness in papillary thyroid cancer (PTC) including PMCs and to lay out the scientific basis for their translation into patient management. In this study we will perform specially designed diffusion weighted MRI (DW-MRI) and dynamic contrast agent MRI (DCE-MRI) protocols in the PTC patients.

DW-MRI allows for quantifying water diffusion which has been shown to be related to tumor cellularity (29). Particularly, appropriate modeling with DW-MRI data acquired at multiple b values will enable quantifying tumor cellularity and vascularity simultaneously (30-32). DCE-MRI with proper compartmental modeling will yield metrics related to tumor-vessel permeability, tumor perfusion, and extracellular-extravascular volume fraction (33, 34). These facts provide the potential of DW-MRI and DCE-MRI metrics as quantitative imaging biomarkers of tumor aggressiveness in PTCs. The DW-MRI and DCE-MRI may ultimately help in personalized management approach, in which imaging biomarkers may be used to recommend either immediate surgery or active surveillance for PTC patients.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven Papillary Thyroid Cancer (regardless of genotype and including all subtypes such as follicular or mixed papillary follicular) or suspicious for Thyroid Cancer
* Thyroidectomy or lobectomy planned as definitive treatment for Thyroid Cancer or patients on active surveillance management approach
* Age ≥18 years

Exclusion Criteria:

* Patient would require anesthesia for the study
* Patients who are claustrophobic Patients with tumor size greater than 5 cm in diameter as measured at imaging (ultrasonography or MRI) before treatment
* Patients who have presence of a known contraindication to MRI

  * Pacemaker
  * Aneurysmal clips
  * Metal implants in field of view
  * Pregnant
  * Age and mental status wherein he/she is unable to cooperate for MRI study Patients who have presence of a known contraindication to DCE-MRI may not participate in that portion of the study
  * Known reaction to Gd-DTPA, contrast agent
  * Chronic kidney disease
  * nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical Head and Neck Cancer clinic MSKCC
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
feasibility of MRI biomarkers | up to six months
  The long-term goal of this work will be to perform clinical trials of personalized management approach, in which imaging biomarkers are used to recommend either immediate surgery or active surveillance for PTC patients.

CONTACTS AND LOCATIONS:
Overall Officials: Amita Dave, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT02178345/ICF_000.pdf